CLINICAL TRIAL: NCT06505122
Title: A Pilot Randomized Controlled Trial (RCT) of a Dyadic Life Review Intervention for Older Patients With Advanced Cancer) and Their Caregivers
Brief Title: Dyadic Life Review Intervention for Older Patients With Advanced Cancer) and Their Caregivers
Acronym: DLR RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Lee Kehoe, PhD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC24051
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Older Adults; Geriatric Oncology; Caregivers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic Life Review (Experimental): The Dyadic Life Review Arm (DLR) consists of 8 sessions delivered by a trained licensed clinician. Each session facilitates a recall of each phase of life. The patient and caregiver will each be asked structured questions to prompt reminiscence of memories from that phase of life. Interventionists are able to use clinical judgment to prompt further or ask follow-up questions or reflections. Additionally, the patient and caregiver will be asked to respond to the other dyad member's memory or reflection. Each session will have flexibility for clinical judgement.
  Interventions: Behavioral: Dyadic Life Review
- Case-As-Usual (No Intervention): The Care-As-Usual (CAU) arm will follow current practices for responding to patient distress. The CAU for patients involves a supportive follow-up phone call from the social work team to further assess the patient's experience of distress. In some instances, the social worker will use their clinical judgement to further refer the patient to community resources to support distress. The number of phone calls and any subsequent community referrals or appointments related to distress that occur will be tracked.

INTERVENTIONS:
Behavioral: Dyadic Life Review — DLR is an intervention that will promote relationship closeness, communication, and psychological distress in both older adults and caregivers.
  Other Names: DLR
  Arms: Dyadic Life Review

SUMMARY:
The purpose of this study is to test the feasibility of a pilot Randomized Controlled Trial (RCT) comparing Dyadic Life Review (DLR) intervention in older adults with advanced cancer and their caregivers to Care-as-Usual (CAU) group, which involves a referral to social work.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility of a pilot Randomized Controlled Trial (RCT) comparing Dyadic Life Review (DLR) intervention in older adults with advanced cancer and their caregivers to Care-as-Usual (CAU) group, which involves a referral to social work. The study will enroll dyads (pairs) of caregivers and older patients with advanced cancer and dyads of caregivers and patients with advanced cancer. A previous single-arm study was performed testing the feasibility of the adapted DLR intervention in older adults with advanced cancer and their caregivers. The single-arm pilot demonstrated DLR was feasible and acceptable by both patients and caregivers. This innovative pilot study will gather data to test the feasibility of a pilot and examine pre-post intervention changes in caregiver psychological distress.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age ≥ 65
* Patient has a Stage III or IV advanced cancer diagnosis of any type
* Score of 4 or more on National Comprehensive Cancer Network (NCCN) Distress Thermometer (DT)*
* Able to read and understand English

Patient Exclusion Criteria:

• Unable to identify caregiver to participate in study

Caregiver Inclusion Criteria:

* One caregiver must enroll with each patient for either subject to be eligible.
* Caregivers will be selected by the patient when asked if there is a "significant other, spouse, romantic partner, or adult child with whom you discuss or can be helpful in health-related matters;"
* Age 50 or older
* Able to reach and understand English

Caregiver Exclusion Criteria:

• Caregivers unable to provide consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
DLR Intervention Enrollment Rate | 18 weeks
  Evaluate the feasibility of DLR in older patients and caregivers based on enrollment rate.
DLR Intervention Retention Rate | 18 weeks
  Evaluate the feasibility of DLR in older patients and caregivers based on retention rate.

SECONDARY OUTCOMES:
Unidimensional Relationship Closeness Scale | 18 weeks
  Quality of relationship with care-receiver: assesses quality of relationship between participant and family member and has demonstrated valid scores across several relationship types, including spouses and other family members. This is a 12-item scale, rated from 1-7 (1=strongly agree, 7=strongly disagree), with a possible total of 84; a higher score indicates a higher level of closeness.
Communication Satisfaction Scale | 18 weeks
  The observation of each partner's level of satisfaction with various aspects of their communication. This is a 12-item scale, rated from 1-5 (1=not at all satisfied, 5=extremely satisfied), with a possible total of 60; a higher score indicates greater satisfaction with communication.
Distress Thermometer | 18 weeks
  A self-report measure to capture distress and identify a list of sources of that distress. This is a 10-item scale, rated from 0-10 (0=no distress, 10=severe distress), with a possible total of 10; a higher score indicates greater distress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No